CLINICAL TRIAL: NCT05131568
Title: Efficacy of a Thermal Insulation System in Inadvertent Hypothermia and Perioperative Comfort
Brief Title: Thermal Insulation System in Inadvertent Hypothermia
Acronym: SIT-3c
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SIT-3c
Record Dates: First submitted 2018-10-18; First posted 2021-11-23 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2018-09

CONDITIONS: Perioperative Hypothermia
Keywords: perioperative hypothermia; thermal insulation; perioperative comfort

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thermal insulation system (Experimental): experimental: layered thermal insulation system
  The system was applied in the upper body to the entrance of the operating room and remained until the exit of the same room.
  The test included the evaluation of temperature, tremors and the visual perception of thermal comfort in 6 moments (T1 - reference temperature - at the entrance of the anesthetic induction room, T2 - at the entrance to the operating room, T3, T4 and T5 - fifteen , thirty and forty-five minutes after the start of surgery, and T6 - leaving the operating room)
  Interventions: Device: Layered thermal insulation system
- Forced air active warming (No Intervention): Control: the same procedures as in the experiment group, were carried out in the control group, except for the intervention.

INTERVENTIONS:
Device: Layered thermal insulation system — No other intervention
  Arms: Thermal insulation system

SUMMARY:
This study compares the effectiveness of a new layered thermal insulation system (SIT-3c) versus the traditional thermal body protection (warmed forced air system) for patients under total knee arthroplasty, during the intra-operative phase.

DETAILED DESCRIPTION:
Protecting patients from the cold in the operating room is a complex problem that has encouraged the search for better and more effective thermal protection systems. Some disadvantages have been observed in the daily use of the recommended thermal protection system (forced warm air).

This study intends to design and evaluate the effectiveness of a three-layer thermal insulation system, comparing its effect with the forced warm air system on temperature variation, shivering incidence and comfort perception, in patients undergoing total knee arthroplasty under neuro-axial anesthesia, during the intra-operative phase.

Participants are randomly assigned to the experimental group (EG) or control group (CG). The experimental group receives as a skin protection the three-layer thermal insulation system (SIT-3c) and the control group receives the usual recommended system (forced warm air).

Both systems are placed at the entrance to the operating room and held on patients during the entire intra-operative phase.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years, with the diagnosis of gonarthrosis, to undergo total elective knee arthroplasty, under neuroaxial anesthesia, who agreed to participate in the study.

Exclusion Criteria:

* With hypothermia or hyperthermia, scheduled for general anesthesia, pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Changes in tympanic temperature (T1) | Baseline (entrance in the operating room)
  Method of assessment - the TTS-400 thermometer, Smiths Medical was used
Changes in tympanic temperature (T2) | immediately after anesthesia
  Method of assessment - the TTS-400 thermometer, Smiths Medical was used
Changes in tympanic temperature (T3) | 15 minutes after beginning surgery
  Method of assessment - the TTS-400 thermometer, Smiths Medical was used
Changes in tympanic temperature (T4) | 30 minutes after beginning surgery
  Method of assessment - the TTS-400 thermometer, Smiths Medical was used
Changes in tympanic temperature (T5) | 45 minutes after beginning surgery
  Method of assessment - the TTS-400 thermometer, Smiths Medical was used
Changes in tympanic temperature (T6) | Up to 10 min after the end of surgery (living the operating room)
  Method of assessment - the TTS-400 thermometer, Smiths Medical was used
Changes in shivering (T1) | Baseline (entrance in the operating room)
  Method of assessment - the Leslie and Sessler Scale, which measures tremors at three levels (0 - no tremors; 1 - slight tremors; 2 - vigorous tremors).
Changes in shivering (T2) | immediately after anesthesia
  Method of assessment - the Leslie and Sessler Scale, which measures tremors at three levels (0 - no tremors; 1 - slight tremors; 2 - vigorous tremors).
Changes in shivering (T3) | 15 minutes after beginning surgery
  Method of assessment - the Leslie and Sessler Scale, which measures tremors at three levels (0 - no tremors; 1 - slight tremors; 2 - vigorous tremors).
Changes in shivering (T4) | 30 minutes after beginning surgery
  Method of assessment - the Leslie and Sessler Scale, which measures tremors at three levels (0 - no tremors; 1 - slight tremors; 2 - vigorous tremors).
Changes in shivering (T5) | 45 minutes after beginning surgery
  Method of assessment - the Leslie and Sessler Scale, which measures tremors at three levels (0 - no tremors; 1 - slight tremors; 2 - vigorous tremors).
Changes in shivering (T6) | Up to 10 min after the end of surgery (living the operating room)
  Method of assessment - the Leslie and Sessler Scale, which measures tremors at three levels (0 - no tremors; 1 - slight tremors; 2 - vigorous tremors).
Changes in visual perception of Thermal comfort (T1) | Baseline (entrance in the operating room)
  Method of assessment - the Visual Comfort Scale, which measures the perception of thermal comfort in two components: numerical (1 to 10) and visual (5 faces). The numerical component varies between 0 (very cold) and 10 (very hot), the value of the thermal neutrality, which means thermal comfort, identified in point 5; and the visual component where five expressive faces are presented. The first one, located between the numbers 0-2, shows strong cold discomfort, the second, located between 2-4, expressed cold discomfort, the third, located in the area of the number 5, expresses a sensation of thermal comfort, the fourth, located between the numbers 6-8, reveals heat discomfort and the fifth, located between 8-10, shows strong heat discomfort.
Changes in visual perception of Thermal comfort (T2) | immediately after anesthesia
  Method of assessment - the Visual Comfort Scale, which measures the perception of thermal comfort in two components: numerical (1 to 10) and visual (5 faces). The numerical component varies between 0 (very cold) and 10 (very hot), the value of the thermal neutrality, which means thermal comfort, identified in point 5; and the visual component where five expressive faces are presented. The first one, located between the numbers 0-2, shows strong cold discomfort, the second, located between 2-4, expressed cold discomfort, the third, located in the area of the number 5, expresses a sensation of thermal comfort, the fourth, located between the numbers 6-8, reveals heat discomfort and the fifth, located between 8-10, shows strong heat discomfort.
Changes in visual perception of Thermal comfort (T3) | 15 minutes after beginning surgery
  Method of assessment - the Visual Comfort Scale, which measures the perception of thermal comfort in two components: numerical (1 to 10) and visual (5 faces). The numerical component varies between 0 (very cold) and 10 (very hot), the value of the thermal neutrality, which means thermal comfort, identified in point 5; and the visual component where five expressive faces are presented. The first one, located between the numbers 0-2, shows strong cold discomfort, the second, located between 2-4, expressed cold discomfort, the third, located in the area of the number 5, expresses a sensation of thermal comfort, the fourth, located between the numbers 6-8, reveals heat discomfort and the fifth, located between 8-10, shows strong heat discomfort.
Changes in visual perception of Thermal comfort (T4) | 30 minutes after beginning surgery
  Method of assessment - the Visual Comfort Scale, which measures the perception of thermal comfort in two components: numerical (1 to 10) and visual (5 faces). The numerical component varies between 0 (very cold) and 10 (very hot), the value of the thermal neutrality, which means thermal comfort, identified in point 5; and the visual component where five expressive faces are presented. The first one, located between the numbers 0-2, shows strong cold discomfort, the second, located between 2-4, expressed cold discomfort, the third, located in the area of the number 5, expresses a sensation of thermal comfort, the fourth, located between the numbers 6-8, reveals heat discomfort and the fifth, located between 8-10, shows strong heat discomfort.
Changes in visual perception of Thermal comfort (T5) | 45 minutes after beginning surgery
  Method of assessment - the Visual Comfort Scale, which measures the perception of thermal comfort in two components: numerical (1 to 10) and visual (5 faces). The numerical component varies between 0 (very cold) and 10 (very hot), the value of the thermal neutrality, which means thermal comfort, identified in point 5; and the visual component where five expressive faces are presented. The first one, located between the numbers 0-2, shows strong cold discomfort, the second, located between 2-4, expressed cold discomfort, the third, located in the area of the number 5, expresses a sensation of thermal comfort, the fourth, located between the numbers 6-8, reveals heat discomfort and the fifth, located between 8-10, shows strong heat discomfort.
Changes in visual perception of Thermal comfort (T6) | Up to 10 min after the end of surgery (living the operating room)
  Method of assessment - the Visual Comfort Scale, which measures the perception of thermal comfort in two components: numerical (1 to 10) and visual (5 faces). The numerical component varies between 0 (very cold) and 10 (very hot), the value of the thermal neutrality, which means thermal comfort, identified in point 5; and the visual component where five expressive faces are presented. The first one, located between the numbers 0-2, shows strong cold discomfort, the second, located between 2-4, expressed cold discomfort, the third, located in the area of the number 5, expresses a sensation of thermal comfort, the fourth, located between the numbers 6-8, reveals heat discomfort and the fifth, located between 8-10, shows strong heat discomfort.

SECONDARY OUTCOMES:
General intraoperative comfort | 30 minutes after beginning surgery
  Method of assessment - the Perioperative Comfort Scale, based on Kolcaba´s theory, composed of 15 items answered by a six-point Likert scale ranging from 1 (totally disagree) to 6 (I totally agree), which measures general aspects of comfort in three dimensions: relief, ease and transcendence.
Thermal intraoperative comfort | 30 minutes after beginning surgery
  Method of assessment - the Thermal Comfort Scale, composed of 9 items answered by a six-point Likert scale ranging from 1 (totally disagree) to 6 (I totally agree), which measures thermal aspects of comfort in two dimensions: physical and emotional.
Ergonomic comfort | 30 minutes after beginning surgery
  Method of assessment - the Ergonomic questionnaire, composed of 10 items answered by a five-point Likert scale ranging from 1 (not at all comfortable) to 5 (very comfortable).

CONTACTS AND LOCATIONS:
Overall Officials: Isaura Carvalho, Dr., Principal Investigator — Hospital of Prelada - Porto
Locations (1):
- University of Porto - Biomedical Sciences Institut, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] AORN Recommended Practices Committee. Recommended practices for the prevention of unplanned perioperative hypothermia. AORN J. 2007 May;85(5):972-4, 976-84, 986-8. doi: 10.1016/j.aorn.2007.04.015. No abstract available. PMID 17533677
- [Background] Fallis WM, Hamelin K, Symonds J, Wang X. Maternal and newborn outcomes related to maternal warming during cesarean delivery. J Obstet Gynecol Neonatal Nurs. 2006 May-Jun;35(3):324-31. doi: 10.1111/j.1552-6909.2006.00052.x. PMID 16700681
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Frank SM, El-Rahmany HK, Cattaneo CG, Barnes RA. Predictors of hypothermia during spinal anesthesia. Anesthesiology. 2000 May;92(5):1330-4. doi: 10.1097/00000542-200005000-00022. PMID 10781278
- [Background] Koeter M, Leijtens B, Koeter S. Effect of thermal reflective blanket placement on hypothermia in primary unilateral total hip or knee arthroplasty. J Perianesth Nurs. 2013 Dec;28(6):347-52. doi: 10.1016/j.jopan.2012.08.007. PMID 24267622
- [Background] Kurz A, Sessler DI, Narzt E, Lenhardt R, Lackner F. Morphometric influences on intraoperative core temperature changes. Anesth Analg. 1995 Mar;80(3):562-7. doi: 10.1097/00000539-199503000-00023. PMID 7864426
- [Background] Morris RH, Wilkey BR. The effects of ambient temperature on patient temperature during surgery not involving body cavities. Anesthesiology. 1970 Feb;32(2):102-7. doi: 10.1097/00000542-197002000-00003. No abstract available. PMID 5414287
- [Background] National Collaborating Centre for Nursing and Supportive Care (UK). The Management of Inadvertent Perioperative Hypothermia in Adults [Internet]. London: Royal College of Nursing (UK); 2008 Apr. Available from http://www.ncbi.nlm.nih.gov/books/NBK53797/ PMID 21678626
- [Background] Shaw CA, Steelman VM, DeBerg J, Schweizer ML. Effectiveness of active and passive warming for the prevention of inadvertent hypothermia in patients receiving neuraxial anesthesia: A systematic review and meta-analysis of randomized controlled trials. J Clin Anesth. 2017 May;38:93-104. doi: 10.1016/j.jclinane.2017.01.005. Epub 2017 Jan 31. PMID 28372696
- [Background] Tramontini CC, Graziano KU. Hypothermia control in elderly surgical patients in the intraoperative period: evaluation of two nursing interventions. Rev Lat Am Enfermagem. 2007 Jul-Aug;15(4):626-31. doi: 10.1590/s0104-11692007000400016. PMID 17923980
- [Background] Welch TC. AANA journal course. Update for nurse anesthetists. A common sense approach to hypothermia. AANA J. 2002 Jun;70(3):227-31. PMID 12078471
- [Background] Hooper VD, Chard R, Clifford T, Fetzer S, Fossum S, Godden B, Martinez EA, Noble KA, O'Brien D, Odom-Forren J, Peterson C, Ross J, Wilson L; ASPAN. ASPAN's evidence-based clinical practice guideline for the promotion of perioperative normothermia: second edition. J Perianesth Nurs. 2010 Dec;25(6):346-65. doi: 10.1016/j.jopan.2010.10.006. No abstract available. PMID 21126665
- See also: 1. Biazzotto, C. B., Brudniewski, M., Schmidt, A. P., & Júnior, J. O. (2006). Hipotermia no Período Peri-Operatório. Rev Bras Anestesiol, 56(1), pp. 89-106. — http://www.scielo.br/pdf/rba/v56n1/v56n1a12.pdf
- See also: Ferreira, J. C., & Patino, C. M. (2016). Randomização: mais do que o lançamento de uma moeda. J Bras Pneumol, 42(5), pp. 310-310. — http://dx.doi.org/10.1590/S1806-37562016000000296
- See also: Insler, S., & Sessler, D. (2006). Perioperative Thermoregulation and Temperature Monitoring. Anesth Clinic, 24, pp. 823-837. — http://doi.org/10.1016/j.atc.2006.09.001